CLINICAL TRIAL: NCT05205239
Title: Intestinal Dysmotility in Patients With Functional Digestive Symptoms
Brief Title: Small Bowel Motility in Patients With Systemic Sclerosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PR(AG)56/2018C
Record Dates: First submitted 2022-01-11; First posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-10

CONDITIONS: System Sclerosis
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Systemic sclerosis (Experimental)
  Interventions: Diagnostic Test: Endoluminal image analysis by capsule endoscopy

INTERVENTIONS:
Diagnostic Test: Endoluminal image analysis by capsule endoscopy — Studies will be performed after discontinuation of medications that could affect gastrointestinal motility for at least 48 hours and overnight fast. Endoluminal images were obtained with the Pillcam capsule (Pillcam SB3 video capsule; Medtronic). Images will be obtained at a fixed 2 per second rate and recorded for a total of 8 hours with the subjects lying comfortably on a hospital bed and the trunk raised 30° above horizontal. Forty-five minutes after gastric exit, participants will be instructed to ingest a liquid meal (Ensure HN; Abbott; 300 mL,1 Kcal/mL). Endoluminal images of the small bowel will be analyzed with a computer program specifically developed in our laboratory for the evaluation of intestinal motility. This previously validated program is based on computer vision techniques, which allow the detection and quantification of contractile and non-contractile patterns characterizing small bowel motility.

SUMMARY:
Several studies using intestinal manometry have reported alterations in small bowel motility in patients with systemic sclerosis. Our aim is to apply endoluminal image analysis to stratify the intestinal motor dysfunction in these patients can be assessed by non-invasive techniques. Consecutive patients with systemic sclerosis referred to our institution will be prospectively investigated using automated non-invasive techniques developed in our laboratory. Intraluminal images of the gut were obtained by capsule endoscopy. Endoluminal image analysis will be performed with original, previously validated programs based on computer vision and machine learning techniques.

ELIGIBILITY:
Inclusion Criteria:

* Systemic sclerosis diagnosed by ACR criteria

Exclusion Criteria:

* Lung transplantation
* End stage kidney disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Motility index score | 8 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Vall d'Hebron, Barcelona, Spain

REFERENCES:
- [Background] Malagelada C, Drozdzal M, Segui S, Mendez S, Vitria J, Radeva P, Santos J, Accarino A, Malagelada JR, Azpiroz F. Classification of functional bowel disorders by objective physiological criteria based on endoluminal image analysis. Am J Physiol Gastrointest Liver Physiol. 2015 Sep 15;309(6):G413-9. doi: 10.1152/ajpgi.00193.2015. Epub 2015 Aug 6. PMID 26251472
- [Background] Segui S, Drozdzal M, Pascual G, Radeva P, Malagelada C, Azpiroz F, Vitria J. Generic feature learning for wireless capsule endoscopy analysis. Comput Biol Med. 2016 Dec 1;79:163-172. doi: 10.1016/j.compbiomed.2016.10.011. Epub 2016 Oct 19. PMID 27810622
- [Background] Malagelada C, Bendezu RA, Segui S, Vitria J, Merino X, Nieto A, Sihuay D, Accarino A, Molero X, Azpiroz F. Motor dysfunction of the gut in cystic fibrosis. Neurogastroenterol Motil. 2020 Sep;32(9):e13883. doi: 10.1111/nmo.13883. Epub 2020 May 31. PMID 32475007